CLINICAL TRIAL: NCT03442959
Title: Resection of the Primary Tumor vs no Resection in Asymptomatic Patients With Unresectable Synchronous Liver Metastases From siNEN
Acronym: SI-NET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO17142
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-02

CONDITIONS: Small Intestinal Neuroendocrine Tumor
Keywords: Small intestine neuroendocrine tumor; palliative surgery
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with primary resection of the Small Intestinal TNE
  Interventions: Other: Data record
- patient without primary resection of the Small Intestinal TNE
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record — characteristics of patients, initial clinical presentation of TNE, management of TNE (primary tumor resection or conservative strategy), five years follow up (locoregional recurrence, complication due to the surgery, complications related to the conservative strategy, death)

SUMMARY:
Small Intestinal neuroendocrine Tumors (SiNETs) incidence is rising. Most of siNETs primaries are localized in jejunum/ileum. At the diagnosis, 50-70% of them present either lymph node (LN) and/or liver metastases (LM). It is admitted that almost 30% of the patients present or will present primary complications. Primary complications include endoluminal obstruction and/or LN-fibrotic mesenteritis with occlusive symptoms, and less frequently haemorrhage and/or intestinal ischemia.However, it is not clear weather this affects patient with or without multiple liver metastases (LM). In this regard, many centres propose to perform primary resection even in patients presenting unresectable LM. Thus, systemic reviews suggest a possible benefit of the primary midgut siNETs resection even in patients with unresectable LM, there is no prospective randomized trial showing the benefit of primary resection in such patients especially those who are totally asymptomatic. Indeed, all retrospective published series have several limitations and the results should be therefore considered with caution.

Theoretical impact of "preventive" resection of midgut primaries in patients with unresectable LM and totally free of occlusive symptoms is controversial. Firstly, it is to avoid primary mechanical complications, and secondly to allow targeting therapeutics to the liver compartment. In this regard, in patients with synchronous unresectable LM from siNENs, ENETS, UKINETS, NANETS guidelines propose, in "a case-by-case" selective approach, the resection of the primary, while NCCN guidelines advocate to do not propose primary resection in such patient if they are free of symptoms with low tumor burden.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Patient with Si-NET and liver metastases considered as non-resectable
* Primary-related "asymptomatic" patient at diagnosis
* Diagnosed during the past 6 months
* No symptoms in relation with the primary or with mesenteric lesions
* Symptoms related to carcinoid syndrome allowed

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosis (in the last 6 months) of asymptomatic primary Si-NET with liver metastases considered as non-resectable between 01/02/2018 and 01/02/2019.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2024-07-03 (Estimated); Study Completion 2025-01-03 (Estimated)

PRIMARY OUTCOMES:
Death | 5 years
  Death due to Small Intestinal neuroendocrine Tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France